CLINICAL TRIAL: NCT02921412
Title: Performance of Fanfilcon A Toric Lenses After at Least One Month Wearing Enfilcon A Toric Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-67
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- enfilcon A (habitual) (No Intervention): All participants wear enfilcon A toric lens (habitual) and then refitted with fanfilcon A toric lenses.
- fanfilcon A (Active Comparator): All participants wear enfilcon A toric lens (habitual) and then refitted with fanfilcon A toric lenses.
  Interventions: Device: fanfilcon A

INTERVENTIONS:
Device: fanfilcon A — contact lens
  Arms: fanfilcon A

SUMMARY:
This is a prospective, multi-center, subject-masked, bilateral, daily wear, two-month dispensing study

DETAILED DESCRIPTION:
The aim of this study is to determine if adapted contact lens wearers enfilcon A toric lenses can be confidently refit into fanfilcon A toric lenses and can be successful after one month of daily wear.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported eye exam in the last two years
* Is a habitual soft toric lens wearer
* Can be successfully fit with study lenses (≥ grade 2 fit acceptance)
* Has a contact lens spherical prescription between -1.00 to -6.00D with a cylinder between -0.75 and -1.75D (Diopters) (inclusive)
* Has a spectacle cylinder of at least 0.75D in each eye.
* Can achieve best corrected spectacle refraction distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Has a contact lens refraction that fits within the available parameters of the study lenses
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so)
* Is willing to comply with the visit schedule.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Has a history of not achieving comfortable CL (Contact Lens) wear (5 days per week; > 8 hours/day)
* Presents with clinically significant anterior segment abnormalities
* Presents with ocular or systemic disease or need of medications which might interfere with contact lens wear
* Presents with slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Significant pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Anterior uveitis or iritis (or history in past year)
  * Seborrheic eczema of eyelid region, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.
* Is frequently using rewetting/ lubricating eye drops (more than once per day)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hospital Contact Lens Service, Miami, Florida
  - Debbie Kim, Closter, New Jersey
  - West Village Eyecare, New York, New York
  - Spokane Eye Clinic, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants were initially enrolled (assigned a study ID), with 1 failing the screening. A total of 36 participants wore the control lens (enfilcon A toric) first and then refitted and dispensed the test lenses (fanfilcon A toric) at baseline visit. There were no discontinuations.
Groups:
- All Participants (Enfilcon A Toric / Fanfilcon A Toric Lenses): All participants wore enfilcon A toric lens (habitual) and then wore fanfilcon A toric lenses for 1 month.
Period: Overall Study
Arm/Group | All Participants (Enfilcon A Toric / Fanfilcon A Toric Lenses)
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed prior to one participant completing the 2 week and 1 month visits.
Groups:
- Enfilcon A Toric / Fanfilcon A Toric: All participants wear enfilcon A toric lens (habitual) and then refitted with fanfilcon A toric lenses at baseline visit.
Arm/Group | Enfilcon A Toric / Fanfilcon A Toric
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: High contrast distance visual acuity is measured by LogMAR.
Time Frame: baseline, 2 weeks, 1 month
Population: Analysis was performed prior to one participant completing the 2 week and 1 month visits.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Enfilcon A Toric (Baseline); Fanfilcon A Toric (Dispense); Fanfilcon A Toric (2 Weeks); Fanfilcon A Toric (1 Month): All participants wear enfilcon A toric lens (habitual) and then refitted with fanfilcon A toric lenses at baseline visit.
Arm/Group | Enfilcon A Toric (Baseline) | Fanfilcon A Toric (Dispense) | Fanfilcon A Toric (2 Weeks) | Fanfilcon A Toric (1 Month)
Number analyzed (Participants) | 36 | 36 | 35 | 35
logMAR | -0.05 (0.05) | -0.05 (0.05) | -0.05 (0.05) | -0.04 (0.04)

2. Primary Outcome: Centration
Description: Lens centration is assessed (optimum, decentration acceptable, decentration unacceptable).
Time Frame: baseline, 2 weeks, 1 month
Population: Analysis was performed prior to one participant completing the 2 week and 1 month visits.
Measure: Count of Participants; unit: Participants
Groups:
- Enfilcon A Toric (Baseline); Fanfilcon A Toric (Dispense); Fanfilcon A Toric (2 Weeks); Fanfilcon A Toric (1 Month): All participants wear enfilcon A toric lens (for 1 month) and then refitted with fanfilcon A toric lenses at baseline visit.
Arm/Group | Enfilcon A Toric (Baseline) | Fanfilcon A Toric (Dispense) | Fanfilcon A Toric (2 Weeks) | Fanfilcon A Toric (1 Month)
Number analyzed (Participants) | 36 | 36 | 35 | 35
Participants
  Optimum | 34 | 35 | 30 | 33
  Acceptable | 1 | 1 | 5 | 2
  Unacceptable | 1 | 0 | 0 | 0

3. Primary Outcome: Corneal Coverage
Description: Corneal coverage will be assessed (yes/no)
Time Frame: baseline, 2 weeks, 1 month
Population: Analysis was performed prior to one participant completing the 2 week and 1 month visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Enfilcon A Toric (Baseline) | Fanfilcon A Toric (Dispense) | Fanfilcon A Toric (2 Weeks) | Fanfilcon A Toric (1 Month)
Number analyzed (Participants) | 36 | 36 | 35 | 35
Participants
  Yes | 36 | 36 | 35 | 35
  No | 0 | 0 | 0 | 0

4. Primary Outcome: Post-blink Movement
Description: Post-blink lens movement assessed using the following evaluations (0-4): 0=Insufficient, unacceptable, 1=Minimal, acceptable, 2=Optimal, 3=Moderate, acceptable, 4=Excessive, unacceptable)
Time Frame: baseline, 2 weeks, 1 month
Population: Analysis was performed prior to one participant completing the 2 week and 1 month visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enfilcon A Toric (Baseline) | Fanfilcon A Toric (Dispense) | Fanfilcon A Toric (2 Weeks) | Fanfilcon A Toric (1 Month)
Number analyzed (Participants) | 36 | 36 | 35 | 35
units on a scale | 1.83 (0.51) | 1.92 (0.50) | 1.69 (0.47) | 1.86 (0.49)

5. Primary Outcome: Fit Acceptability
Description: Investigator fit acceptability for each lens pair. Scale 0-4: (0=should not be worn, 1=borderline but unacceptable, 2=minimally acceptable, early review, 3=not perfect but OK to dispense, 4=perfect)
Time Frame: baseline, 2 weeks, 1 month
Population: Analysis was performed prior to one participant completing the 2 week and 1 month visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enfilcon A Toric (Baseline) | Fanfilcon A Toric (Dispense) | Fanfilcon A Toric (2 Weeks) | Fanfilcon A Toric (1 Month)
Number analyzed (Participants) | 36 | 36 | 35 | 35
units on a scale | 3.3 (0.6) | 3.3 (0.5) | 3.1 (0.8) | 3.1 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse event data collected at all scheduled visits over a 1 month period of time
Groups:
- All Participants (Enfilcon A Toric / Fanfilcon A Toric Lenses): All participants wore enfilcon A toric lenses (habitual) and then refitted with fanfilcon A toric lenses at baseline visit.
Arm/Group | All Participants (Enfilcon A Toric / Fanfilcon A Toric Lenses)
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any results communications and has ability to review.

DOCUMENTS (2):
  • Informed Consent Form (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT02921412/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02921412/Prot_SAP_002.pdf